CLINICAL TRIAL: NCT01922739
Title: A 6-Month, Open-Label, Extension Study to Evaluate the Safety of Hydrocodone Bitartrate Extended-Release Tablets (CEP-33237) at 15 to 90 mg Every 12 Hours for Relief of Moderate to Severe Pain in Patients With Chronic Low Back Pain Who Require Opioid Treatment for an Extended Period of Time
Brief Title: Open-Label, Extension Study to Evaluate the Safety of Hydrocodone Bitartrate Extended-Release Tablets
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C33237/3104
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Low Back Pain
Keywords: low back pain; hydrocodone bitartrate; opioids
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydrocodone ER (Experimental): Participants were administered hydrocodone ER tablets orally at dosages of 15, 30, 45, 60, or 90 mg every 12 hours at the dosage deemed successful for managing their pain. If enrolled under the original protocol, there was a double-blind titration period of four weeks to adjust the dose taken in study 3103 (NCT01789970). If enrolled under the amended protocol, there was an open-label adjustment period of three weeks to adjust the dose taken in study 3103 (NCT01789970). Both versions of protocol 3104 followed the titration/adjustment period with a open-label treatment period of 22 weeks.
  Interventions: Drug: Hydrocodone ER; Drug: Placebo

INTERVENTIONS:
Drug: Hydrocodone ER — Participants were instructed to take hydrocodone ER tablets orally with a glass of water on an empty stomach at least 1 hour before or 2 hours after eating.
  Other Names: CEP-33237; Hydrocodone bitartrate extended-release tablets
Drug: Placebo — During the double-blind titration period used in the original protocol, placebo tablets matching each dose of hydrocodone bitartrate ER tablets (active drug) were used to maintain the blind but not for purposes of comparison.

SUMMARY:
This is a 6-month, nonrandomized, open-label extension study to assess the long-term safety of hydrocodone bitartrate extended-release (ER) tablets in patients with moderate to severe chronic low back pain who require continuous opioid treatment for an extended period of time.

To be eligible for Study 3104, patients were required to have completed the entire double blind treatment period on study drug (either placebo or hydrocodone bitartrate ER tablets) through week 12 of Study 3103 (NCT01789970) and to have met the entry criteria for Study 3104.

DETAILED DESCRIPTION:
Eligible patients from Study 3103 (NCT01789970) were enrolled for participation in this extension study. For these patients, the final study visit in Study 3103 was visit 1 for this study (also referred to as the titration or adjustment baseline visit, depending on whether the patient was enrolled under the original or amended protocol, respectively). The original protocol was amended after 26 patients had been enrolled in the study. Those who were enrolled under the original protocol participated in a double-blind titration period of up to approximately 4 weeks followed by an open-label treatment period of 22 weeks. Those patients who were enrolled under the amended protocol participated in an open-label adjustment period of up to approximately 3 weeks followed by an open-label treatment period of 22 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have participated in and completed the entire double-blind treatment period on study drug through the final study visit (week 12) of study 3103.

   NOTE: Patients who had a final on-treatment visit (i.e. prior to week 12) are not permitted to participate in study 3104.
2. The patient is able to speak English and is willing to provide written informed consent for study 3104, including re-signing a written opioid agreement, to participate in this study.
3. Women of childbearing potential (not surgically sterile or 2 years postmenopausal) must use a medically accepted method of contraception, agree to continue use of this method for the duration of the study and for 30 days after participation in the study, and have a negative pregnancy test at screening. Acceptable methods of contraception include barrier method with spermicide, intrauterine device (IUD), or steroidal contraceptive (oral, transdermal, implanted, and injected) in conjunction with a barrier method. NOTE: A woman will be considered surgically sterile if she has had a tubal ligation, hysterectomy, bilateral salpingo-oophorectomy or bilateral oophorectomy, or hysterectomy with bilateral salpingo-oophorectomy.
4. The patient must be willing and able to successfully self-administer the study drug, comply with study restrictions, and return to the study center for scheduled study visits, as specified in the protocol.
5. The patient must not participate in any other study involving an investigational agent (excluding those who participated in study 3103) while enrolled in the present study.

Exclusion Criteria:

1. The patient's current source of pain is different from the low back pain the patient was experiencing at entry into study 3103. NOTE: Any additional source of pain for a patient must be discussed with the medical monitor.
2. The patient has current evidence of alcohol or other substance abuse with the exception of nicotine or caffeine.
3. The patient has developed, during study 3103, a medical or psychiatric disease (including suicidality) that, in the opinion of the investigator, would compromise collected data.
4. The patient is expected to have surgery during the study.
5. The patient is pregnant or lactating.
6. The patient has developed an active malignancy (excluding basal cell carcinoma) during study 3103.
7. The patient has known human immunodeficiency virus (HIV).
8. In the judgment of the investigator, the patient has any clinically significant deviation from normal in the physical examination and/or clinical laboratory test values.
9. The patient has developed cardiopulmonary disease that would, in the opinion of the investigator, significantly increase the risk of treatment with opioids.
10. The patient is receiving a monoamine oxidase inhibitor (MAOI).

    * Other exclusion criteria apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (61):
- United States (61):
  - Teva Investigational Site 10412, Birmingham, Alabama
  - Teva Investigational Site 10426, Mobile, Alabama
  - Teva Investigational Site 10436, Montgomery, Alabama
  - Teva Investigational Site 10363, Phoenix, Arizona
  - Teva Investigational Site 10366, Phoenix, Arizona
  - Teva Investigational Site 10437, Tucson, Arizona
  - Teva Investigational Site 10358, Anaheim, California
  - Teva Investigational Site 10408, Bell Gardens, California
  - Teva Investigational Site 10425, Carmichael, California
  - Teva Investigational Site 10390, Cerritos, California
  - Teva Investigational Site 10429, El Cajon, California
  - Teva Investigational Site 10423, Escondido, California
  - Teva Investigational Site 10391, Huntington Park, California
  - Teva Investigational Site 10370, Los Angeles, California
  - Teva Investigational Site 10392, Sherman Oaks, California
  - Teva Investigational Site 10398, Thousand Oaks, California
  - Teva Investigational Site 10428, Torrance, California
  - Teva Investigational Site 10361, Walnut Creek, California
  - Teva Investigational Site 10369, DeLand, Florida
  - Teva Investigational Site 10379, Fort Lauderdale, Florida
  - Teva Investigational Site 10365, Jacksonville, Florida
  - Teva Investigational Site 10445, Leesburg, Florida
  - Teva Investigational Site 10362, Orlando, Florida
  - Teva Investigational Site 10381, Ormond Beach, Florida
  - Teva Investigational Site 10357, Plantation, Florida
  - Teva Investigational Site 10435, Royal Palm Beach, Florida
  - Teva Investigational Site 10432, Columbus, Georgia
  - Teva Investigational Site 10383, Marietta, Georgia
  - Teva Investigational Site 10385, Marietta, Georgia
  - Teva Investigational Site 10444, Newnan, Georgia
  - Teva Investigational Site 10431, Meridian, Idaho
  - Teva Investigational Site 10743, Meridian, Idaho
  - Teva Investigational Site 10411, Chicago, Illinois
  - Teva Investigational Site 10440, Newburgh, Indiana
  - Teva Investigational Site 10419, New Orleans, Louisiana
  - Teva Investigational Site 10359, Shreveport, Louisiana
  - Teva Investigational Site 10389, Fall River, Massachusetts
  - Teva Investigational Site 10388, Bay City, Michigan
  - Teva Investigational Site 10397, Biloxi, Mississippi
  - Teva Investigational Site 10406, Hazelwood, Missouri
  - Teva Investigational Site 10401, St Louis, Missouri
  - Teva Investigational Site 10376, Omaha, Nebraska
  - Teva Investigational Site 10399, Las Vegas, Nevada
  - Teva Investigational Site 10409, Berlin, New Jersey
  - Teva Investigational Site 10439, Buffalo, New York
  - Teva Investigational Site 10410, New York, New York
  - Teva Investigational Site 10414, Winston-Salem, North Carolina
  - Teva Investigational Site 10446, Oklahoma City, Oklahoma
  - Teva Investigational Site 10430, Duncansville, Pennsylvania
  - Teva Investigational Site 10386, Mechanicsburg, Pennsylvania
  - Teva Investigational Site 10373, Tipton, Pennsylvania
  - Teva Investigational Site 10405, Austin, Texas
  - Teva Investigational Site 10364, Dallas, Texas
  - Teva Investigational Site 10372, Dallas, Texas
  - Teva Investigational Site 10371, Houston, Texas
  - Teva Investigational Site 10377, Lake Jackson, Texas
  - Teva Investigational Site 10374, Plano, Texas
  - Teva Investigational Site 10378, San Antonio, Texas
  - Teva Investigational Site 10402, Salt Lake City, Utah
  - Teva Investigational Site 10420, Bellevue, Washington
  - Teva Investigational Site 10433, Everett, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 183 patients with moderate to severe chronic low back pain completed Study 3103 and were screened and eligible for enrollment into this study. One patient chose not to participate prior to enrollment.
Pre-assignment Details: Of the 182 participants who enrolled into Study 3104, 26 participants enrolled under the original protocol and 156 participants enrolled under the amended protocol.
Period: Titration/Adjustment Period
Arm/Group | Hydrocodone ER
Started | 182
Safety Analysis Set | 182
Completed | 170
Not Completed | 12
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 3
Period: Open-label Treatment Period
Arm/Group | Hydrocodone ER
Started | 170
Treatment SAS and FAS | 170 (SAS = safety analysis set FAS = full analysis set)
Completed | 136
Not Completed | 34
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 14
Not completed — Noncompliance to study medication | 3
Not completed — Protocol Violation | 5
Not completed — Pregnancy | 1
Not completed — Noncompliance to study procedures | 1
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 1
Not completed — Sponsor request - investigator leaving | 1

BASELINE CHARACTERISTICS:
Population: Enrolled participants
Groups:
- Hydrocodone ER - Opioid Naive: Participants were administered hydrocodone ER tablets at dosages of 15, 30, 45, 60, or 90 mg every 12 hours at the dosage deemed successful for managing their pain. Opioid-naïve participants were defined as those who were taking tramadol or less than 10 mg per day of oxycodone, or equivalent (including around-the-clock and rescue medication) for the 14 days before screening in the C33237/3103 (NCT01789970) study.
- Hydrocodone ER - Opioid Experienced: Participants were administered hydrocodone ER tablets at dosages of 15, 30, 45, 60, or 90 mg every 12 hours at the dosage deemed successful for managing their pain. Opioid-experienced participants were defined as those who were taking 10 mg or more per day of oxycodone, or equivalent (including around-the-clock and rescue medication) for the 14 days before screening in the C33237/3103 (NCT01789970) study.
- Total: Total of all reporting groups
Arm/Group | Hydrocodone ER - Opioid Naive | Hydrocodone ER - Opioid Experienced | Total
Number analyzed (Participants) | 109 | 73 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (13.30) | 55.8 (12.37) | 52.3 (13.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 40 | 100
  Male | 49 | 33 | 82
Age Group [Count of Participants; unit: Participants]
  <=65 years | 94 | 53 | 147
  >65 years | 15 | 20 | 35
Race [Count of Participants; unit: Participants]
  White | 69 | 58 | 127
  Black | 27 | 12 | 39
  Asian | 9 | 1 | 10
  American Indian or Alaskan Native | 2 | 1 | 3
  Pacific Islander | 1 | 0 | 1
  Other | 1 | 1 | 2
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 4 | 28
  Non-Hispanic and non-Latino | 85 | 69 | 154
Weight [Mean (Standard Deviation); unit: kg] | 94.2 (24.56) | 94.2 (25.07) | 94.2 (24.69)
Height [Mean (Standard Deviation); unit: cm] | 169.3 (10.77) | 172.1 (11.18) | 170.4 (10.99)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.9 (8.41) | 31.8 (8.27) | 32.5 (8.35)
Duration Since Diagnosis of Chronic Low Back Pain [Mean (Standard Deviation); unit: years] — Relative to the start of study 3101
  years | 10.7 (10.33) | 12.8 (11.43) | 11.6 (10.80)
Duration on Opioid Therapy [Mean (Standard Deviation); unit: years] | 2.1 (4.72) | 4.8 (4.06) | 3.2 (4.65)
Worst Pain Intensity (WPI) Score [Mean (Standard Deviation); unit: units on a scale] — The WPI was recorded daily by participants in an electronic diary using an 11-point numerical rating scale (NRS-11), a Likert-type scale in which 0=no pain and 10=the worst pain imaginable. Participants selected the number that best described their worst pain intensity over the last 24 hours.
  170 representing participants in the Full Analysis Set which includes participants who had at least one post-baseline efficacy assessment. The timeframe for this measurement is the start of the Open-Label Treatment Period. See outcome #7 for change from baseline values. Population: for some individual participants, the data values were missing
  units on a scale
    number analyzed (Participants) | 106 | 64 | 170
    (all) | 3.7 (1.71) | 4.6 (2.13) | 4.1 (1.92)
Average Pain Intensity (API) [Mean (Standard Deviation); unit: units on a scale] — Measure Description: The API was recorded daily by participants in an electronic diary using an 11-point numerical rating scale (NRS-11), a Likert-type scale in which 0=no pain and 10=the worst pain imaginable. Participants selected the number that best described their average pain intensity over the last 24 hours.
  170 representing participants in the Full Analysis Set which includes participants who had at least one post-baseline efficacy assessment. The timeframe for this measurement is the start of the Open-Label Treatment Period. See outcome #8 for change from baseline values. Population: for some individual participants, the data value was missing
  units on a scale
    number analyzed (Participants) | 106 | 64 | 170
    (all) | 2.6 (1.41) | 3.0 (1.78) | 2.7 (1.57)

OUTCOME MEASURES:

1. Primary Outcome: Participants With Adverse Events
Description: An adverse event (AE) was defined in the protocol as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an inability to carry out usual activities. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 of the Titration/Adjustment Period to Week 22 of the Treatment Period (total of 25-26 weeks)
Population: Safety Analysis Set for the Titration/Adjustment period; Post-Titration/Post-Adjustment Safety Analysis Set for the Open-Label Treatment Period
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Double-Blind Titration Period: Participants were administered hydrocodone ER tablets orally at dosages of 15, 30, 45, 60, or 90 mg every 12 hours at the dosage deemed successful for managing their pain.
  As defined in the original protocol, participants who received placebo during the double-blind treatment period in Study 3103 took hydrocodone bitartrate ER tablets (and matching placebo) every 12 hours titrated to an effective dosage over approximately 4 weeks.
- Hydrocodone ER: Double-Blind Titration Period: Participants were administered hydrocodone ER tablets orally at dosages of 15, 30, 45, 60, or 90 mg every 12 hours at the dosage deemed successful for managing their pain.
  As defined in the original protocol, participants who received hydrocodone ER during the double-blind treatment period in Study 3103 took hydrocodone ER tablets and matching placebo every 12 hours titrated to an effective dosage over approximately 4 weeks.
- Placebo: Open-Label Adjustment Period: Participants were administered hydrocodone ER tablets orally at dosages of 15, 30, 45, 60, or 90 mg every 12 hours at the dosage deemed successful for managing their pain.
  As defined in the amended protocol, participants who received placebo during the double-blind treatment period in Study 3103 took hydrocodone ER every 12 hours titrated to an effective dosage over approximately 3 weeks.
- Hydrocodone ER: Open-Label Adjustment Period: Participants were administered hydrocodone ER tablets orally at dosages of 15, 30, 45, 60, or 90 mg every 12 hours at the dosage deemed successful for managing their pain.
  As defined in the amended protocol, participants who received hydrocodone ER during the double-blind treatment period in Study 3103 took hydrocodone ER every 12 hours titrated to an effective dosage over approximately 3 weeks.
- Hydrocodone ER: Open-Label Treatment Period: Participants were administered hydrocodone ER tablets at dosages of 15, 30, 45, 60, or 90 mg every 12 hours at the dosage deemed successful during the Titration/Adjustment period for managing their pain. The Open-Label Treatment Period lasted 22 weeks.
Arm/Group | Placebo: Double-Blind Titration Period | Hydrocodone ER: Double-Blind Titration Period | Placebo: Open-Label Adjustment Period | Hydrocodone ER: Open-Label Adjustment Period | Hydrocodone ER: Open-Label Treatment Period
Number analyzed (Participants) | 10 | 16 | 68 | 88 | 170
Participants
  Any AE | 4 | 2 | 34 | 25 | 88
  Severe AE | 0 | 0 | 1 | 2 | 11
  Treatment-related AE | 3 | 2 | 21 | 10 | 26
  Deaths | 0 | 0 | 0 | 0 | 0
  Serious AE | 0 | 0 | 0 | 1 | 10
  Withdrawals from treatment due to AE | 1 | 0 | 2 | 1 | 5

2. Primary Outcome: Participants With Potentially Clinically Significant Abnormal Laboratory Values
Description: Data represents participants with potentially clinically significant abnormal serum chemistry, hematology and urinalysis values.
  Significance criteria:
  * Blood urea nitrogen: >=10.71 mmol/L
  * Creatinine: >=177 μmol/L
  * Uric acid: M>=625, F>=506 μmol/L
  * Aspartate aminotransferase (AST): >=3* upper limit of normal (ULN)
  * Alkaline phosphatase: >=3* upper limit of normal (ULN)
  * Gamma-glutamyl transpeptidase (GGT): >=3* upper limit of normal (ULN)
  * Serum white blood cells: >=20 * 10^9/L
  * Hemoglobin: M<=115, F<=95 g/dL
  * Hematocrit: M<0.37, F<0.32 L/L
  * Eosinophils: >=10.0 %
  * Platelets: <=75 * 10^9/L
  * Absolute neutrophils: <=1.0 * 10^9/L
  * Urinalysis: Glucose, Ketones, and Total Protein: >=2 unit increase from baseline
Time Frame: End of trial visit (up to week 22 of Open-label Treatment Period which is up to week 26 including the titration/adjustment period)
Population: The Full Analysis Set includes all participants who took at least one dose of study drug and who had at least 1 post-baseline efficacy assessment. Participants with a post-baseline result for each test are counted as part of the number of participants analyzed for that test.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocodone ER
Number analyzed (Participants) | 170
Participants
  Blood urea nitrogen: number analyzed (Participants) | 160
  Blood urea nitrogen | 5
  Creatinine: number analyzed (Participants) | 160
  Creatinine | 1
  Uric acid: number analyzed (Participants) | 160
  Uric acid | 5
  AST: number analyzed (Participants) | 160
  AST | 1
  Alkaline phosphatase: number analyzed (Participants) | 160
  Alkaline phosphatase | 1
  GGT: number analyzed (Participants) | 160
  GGT | 7
  Serum white blood cells: number analyzed (Participants) | 158
  Serum white blood cells | 1
  Hemoglobin: number analyzed (Participants) | 158
  Hemoglobin | 4
  Hematocrit: number analyzed (Participants) | 158
  Hematocrit | 5
  Eosinophils: number analyzed (Participants) | 158
  Eosinophils | 1
  Platelets: number analyzed (Participants) | 158
  Platelets | 1
  Absolute neutrophils: number analyzed (Participants) | 158
  Absolute neutrophils | 1
  Urine glucose: number analyzed (Participants) | 155
  Urine glucose | 4
  Urine ketones: number analyzed (Participants) | 155
  Urine ketones | 1
  Urine total protein: number analyzed (Participants) | 155
  Urine total protein | 1

3. Primary Outcome: Participants With Potentially Clinically Significant Abnormal Vital Signs Values
Description: Data represents participants with potentially clinically significant (PCS) vital sign values.
  Significance criteria
  * Pulse - high: >=120 and increase of >= 15 beats/minute from baseline
  * Pulse - low: <=50 and decrease of >=15 beats/minute
  * Systolic blood pressure - high: >=180 and increase >=20 mmHg
  * Systolic blood pressure - low: <=90 and decrease >=20 mmHg
  * Diastolic blood pressure - high: >=105 and increase of >=15 mmHg
  * Diastolic blood pressure - low: <=50 and decrease of >=15 mmHg
Time Frame: Day 1 of the Titration/Adjustment Period to Week 22 of the Treatment Period (total of 25-26 weeks)
Population: The Full Analysis Set includes all participants who took at least one dose of study drug and who had at least 1 post-baseline efficacy assessment. Participants with a post-baseline vital sign result are counted as part of the number of participants analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocodone ER
Number analyzed (Participants) | 178
Participants
  Pulse - high | 1
  Pulse - low | 1
  Systolic blood pressure - high | 1
  Systolic blood pressure - low | 3
  Diastolic blood pressure - high | 1
  Diastolic blood pressure - low | 2

4. Primary Outcome: Participants With Shifts From Normal to Abnormal in Physical Examination Findings
Description: The endpoint visit or early termination visit was an abbreviated exam. Endpoint refers to the last observation carried forward.
Time Frame: as for outcome 2
Population: Post-Titration Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocodone ER
Number analyzed (Participants) | 170
Participants
  Normal at baseline - Abnormal at Endpoint | 20
  Abnormal findings reported as adverse events | 7

5. Primary Outcome: Shifts From Baseline to Endpoint (Treatment Period) in Electrocardiogram (ECG) Findings
Description: A 12-lead ECG was conducted at the final visit for study 3103 which is used as baseline for this study, and at week 22 of the treatment period [or early termination]). A qualified physician at the study center was responsible for providing interpretation of the ECG.
  Endpoint refers to the last observation carried forward.
Time Frame: Baseline (final visit for study 3103), End of trial visit (up to week 22 of Open-label Treatment Period which is up to week 26 including the titration/adjustment period)
Population: Post-Titration Safety Analysis Set. Includes participants who have both baseline and endpoint data.
Measure: Count of Participants; unit: Participants
Groups:
- Hydrocodone ER: Participants were administered hydrocodone ER tablets at dosages of 15, 30, 45, 60, or 90 mg every 12 hours at the dosage deemed successful for managing their pain. If enrolled under the original protocol, there was a double-blind titration period of four weeks to adjust the dose taken in study 3103 (NCT01789970). If enrolled under the amended protocol, there was an open-label adjustment period of three weeks to adjust the dose taken in study 3103 (NCT01789970). Both were followed by an open-label treatment period of 22 weeks.
Arm/Group | Hydrocodone ER - Opioid Naive | Hydrocodone ER - Opioid Experienced | Hydrocodone ER
Number analyzed (Participants) | 97 | 60 | 157
Participants
  Baseline normal - Endpoint normal | 26 | 19 | 45
  Baseline normal - Endpoint abnormal | 18 | 11 | 29
  Baseline abnormal - Endpoint normal | 11 | 8 | 19
  Baseline abnormal - Endpoint abnormal | 42 | 22 | 64

6. Primary Outcome: Participants With Clinically Significant (CS) Hearing Changes From Baseline to the Final Visit in Pure Tone Audiometry Test Results
Description: Pure tone audiometry was performed by trained personnel. Hearing loss was classified in degrees of hearing from normal to profound. This classification was determined by the hearing threshold (or the softest sound detected at a specific frequency). The exact ranges that classified hearing loss depended on the exact technique used during testing and on the patient's age. These values were provided by each audiology laboratory that performed the test. For serial audiograms, the criteria for a clinically significant hearing change were based on guidance from the American Speech Language Hearing Association (ASHA 1994, cited in [Konrad-Martin et al 2005]). These criteria included the following: greater than 20 decibels (dB) pure tone threshold shift at 1 frequency; greater than 10 dB shift at 2 consecutive test frequencies; or threshold response shifting to "no response" at 3 consecutive test frequencies.
Time Frame: Baseline was within two weeks of the final study visit in study 3103; during study exam was within two weeks of the end of trial visit for study 3104 (up to study week 26)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocodone ER - Opioid Naive | Hydrocodone ER - Opioid Experienced | Hydrocodone ER
Number analyzed (Participants) | 109 | 73 | 182
Participants | 11 | 7 | 18

7. Secondary Outcome: Change From Baseline to Weeks 2, 6, 10, 14, 18, 22 and Endpoint of the Treatment Period in Daily Worst Pain Intensity (WPI) Scores During the Previous 24 Hours for Each Visit
Description: The WPI was recorded daily by participants in an electronic diary using an 11-point numerical rating scale (NRS-11), a Likert-type scale in which 0=no pain and 10=the worst pain imaginable. At each visit, participants selected the number that best described their worst pain intensity over the last 24 hours. Negative change from baseline scores indicate improvement in pain control.
  Endpoint refers to the last observation carried forward.
Time Frame: Baseline (Day 0 of Treatment Period), Weeks 2, 6, 10, 14, 18, 22 and Endpoint during the Open-Label Treatment Period
Population: Full Analysis Set includes participants who had at least one post-baseline efficacy assessment. Participants contributing to each time point are counted as part of the number of participants analyzed for that test.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Hydrocodone ER - Opioid Experienced: Participants were administered extended-release hydrocodone tablets at dosages of 15, 30, 45, 60, or 90 mg every 12 hours at the dosage deemed successful for managing their pain. Opioid-experienced participants were defined as those who were taking 10 mg or more per day of oxycodone, or equivalent (including around-the-clock and rescue medication) for the 14 days before screening in the C33237/3103 (NCT01789970) study.
- Hydrocodone ER: Participants were administered extended-release hydrocodone tablets at dosages of 15, 30, 45, 60, or 90 mg every 12 hours at the dosage deemed successful for managing their pain. If enrolled under the original protocol, there was a double-blind titration period of four weeks to adjust the dose taken in study 3103 (NCT01789970). If enrolled under the amended protocol, there was an open-label period of three weeks to adjust the dose taken in study 3103 (NCT01789970). Both were followed by an open label treatment period of 22 weeks.
Arm/Group | Hydrocodone ER - Opioid Naive | Hydrocodone ER - Opioid Experienced | Hydrocodone ER
Number analyzed (Participants) | 106 | 64 | 170
units on a scale
  Week 2: number analyzed (Participants) | 105 | 63 | 168
  Week 2 | 0.0 (1.23) | 0.2 (1.28) | 0.1 (1.25)
  Week 6: number analyzed (Participants) | 98 | 63 | 161
  Week 6 | 0.1 (1.63) | 0.1 (1.76) | 0.1 (1.68)
  Week 10): number analyzed (Participants) | 94 | 57 | 151
  Week 10) | 0.0 (1.70) | 0.0 (1.68) | 0.0 (1.69)
  Week 14: number analyzed (Participants) | 90 | 54 | 144
  Week 14 | -0.4 (1.70) | -0.2 (1.82) | -0.3 (1.74)
  Week 18: number analyzed (Participants) | 86 | 53 | 139
  Week 18 | -0.3 (1.73) | -0.4 (1.95) | -0.3 (1.81)
  Week 22: number analyzed (Participants) | 83 | 53 | 136
  Week 22 | -0.1 (1.91) | -0.2 (1.90) | -0.1 (1.90)
  Endpoint | 0.0 (1.87) | 0.1 (1.96) | 0.0 (1.90)

8. Secondary Outcome: Change From Baseline to Weeks 2, 6, 10, 14, 18, 22 and Endpoint of the Treatment Period in Daily Average Pain Intensity (API) Scores During the Previous 24 Hours for Each Visit
Description: The API was recorded daily by participants in an electronic diary using an 11-point numerical rating scale (NRS-11), a Likert-type scale in which 0=no pain and 10=the worst pain imaginable. Participants selected the number that best described their average pain intensity over the last 24 hours. Negative change from baseline scores indicate improvement in pain control.
  Endpoint refers to the last observation carried forward.
Time Frame: Baseline (Day 0 of Treatment Period), Weeks 2, 6, 10, 14, 18, 22 and Endpoint during the Open-Label Treatment Period
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hydrocodone ER - Opioid Naive | Hydrocodone ER - Opioid Experienced | Hydrocodone ER
Number analyzed (Participants) | 106 | 64 | 170
units on a scale
  Week 2: number analyzed (Participants) | 105 | 63 | 168
  Week 2 | -0.1 (0.95) | 0.1 (1.18) | 0.0 (1.05)
  Week 6: number analyzed (Participants) | 98 | 63 | 161
  Week 6 | 0.1 (1.34) | 0.0 (1.52) | 0.1 (1.41)
  Week 10: number analyzed (Participants) | 94 | 57 | 151
  Week 10 | -0.1 (1.45) | -0.1 (1.43) | -0.1 (1.44)
  Week 14: number analyzed (Participants) | 90 | 54 | 144
  Week 14 | -0.3 (1.27) | -0.2 (1.54) | -0.2 (1.37)
  Week 18: number analyzed (Participants) | 86 | 53 | 139
  Week 18 | -0.2 (1.35) | -0.4 (1.57) | -0.3 (1.44)
  Week 22: number analyzed (Participants) | 83 | 53 | 136
  Week 22 | -0.2 (1.54) | -0.3 (2.03) | -0.3 (1.74)
  Endpoint | -0.1 (1.55) | 0.1 (2.20) | 0.0 (1.82)

9. Secondary Outcome: Percentage of Participants Withdrawn From the Study For Lack of Efficacy
Description: Percentage of patients who withdrew from the study for lack of efficacy, as indicated on the early termination form of the case report form (CRF).
Time Frame: Day 1 of the Titration/Adjustment Period to Week 22 of the Treatment Period (total of 25-26 weeks)
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Hydrocodone ER
Number analyzed (Participants) | 182
percentage of participants | 2

ADVERSE EVENTS:
Time Frame: Titration/Adjustment period: Day 1 up to Week 4 Open-label Treatment period: Week 4 to Week 26
Groups:
- Hydrocodone ER - Titration/Adjustment Period: Participants were administered hydrocodone ER tablets at dosages of 15, 30, 45, 60, or 90 mg every 12 hours at the dosage deemed successful for managing their pain. The titration/adjustment period lasted 3-4 weeks.
- Hydrocodone ER - Open-Label Treatment Period: Participants were administered hydrocodone ER tablets at dosages of 15, 30, 45, 60, or 90 mg every 12 hours at the dosage deemed successful during the Titration/Adjustment period for managing their pain. The Treatment Period lasted 22 weeks.
Arm/Group | Hydrocodone ER - Titration/Adjustment Period | Hydrocodone ER - Open-Label Treatment Period
Serious Adverse Events (participants affected / at risk) | 1/182 | 10/170
Other Adverse Events (participants affected / at risk) | 27/182 | 20/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrocodone ER - Titration/Adjustment Period (N=182) | Hydrocodone ER - Open-Label Treatment Period (N=170)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrocodone ER - Titration/Adjustment Period (N=182) | Hydrocodone ER - Open-Label Treatment Period (N=170)
Constipation (Gastrointestinal disorders) | 9 (9) | 12 (13)
Nausea (Gastrointestinal disorders) | 19 (19) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.